CLINICAL TRIAL: NCT05112835
Title: Brolucizumab Treatment Experience Study of Patients With Neovascular Age-related Macular Degeneration (nAMD) in UK Routine Clinical Practice (BESRA)
Brief Title: Brolucizumab Treatment Experience Study of Patients With nAMD in UK Routine Clinical Practice
Acronym: BESRA
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258AGB02
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: brolucizumab intravitreal injections; nAMD; UK
MeSH Terms: interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- brolucizumab: brolucizumab intravitreal injections in patients with nAMD treated in the UK
  Interventions: Other: brolucizumab

INTERVENTIONS:
Other: brolucizumab — There is no treatment allocation. The decision to administer brolucizumab is made by the treating physician independent of the study, prior to the inclusion of the patient into the study

SUMMARY:
BESRA is a national, multi-center, prospective, observational study to assess the effectiveness of brolucizumab intravitreal injections in patients with nAMD treated in the UK.

DETAILED DESCRIPTION:
Data will be collected in a standardized manner from hospital medical records (paper and electronic) at participating centers for up to 60 months post- initiation of brolucizumab. In addition to the collection of data from medical records, retinal OCT images collected during the first two years of treatment will be transferred to a central reading center for independent grading and interpretation, in order to support the validity of anatomical measurements relevant to the primary and secondary study objectives.

Patients will be treated with brolucizumab according to routine clinical practice, independent of the study setting.

Key study design definitions:

* Index date: the date of the first brolucizumab injection.
* Index eye: the first eye to be injected with brolucizumab (analyses will be conducted for the index eye only, unless otherwise stated).
* Post-index period: time between index date and the earliest of treatment discontinuation, date of death or the date of the last recorded visit within the 60 months post-index (2-month window).
* Study period: The period between 01 September 2020 and 01 March 2027, to allow 6 months pre-index period and up to 60 months (±2 months window) follow-up for each enrolled patient.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of nAMD
2. ≥50 years of age at index date
3. Receipt of at least one injection of brolucizumab during the eligibility period
4. Able and willing to provide signed informed consent

Exclusion Criteria:

1. Received treatment for retinal vein occlusion, diabetic macular edema (DME) and/or myopic choroidal neovascularization (mCNV), and/or has received a new diagnosis of diabetes-related macular degeneration in the index eye within 6 months prior to the index date
2. Receipt of anti-VEGF treatment other than brolucizumab in the index eye at index date
3. Any active intraocular or periocular infection or active intraocular inflammation in the index eye at index date
4. Has been on anti-VEGF treatment for longer than 3 years (before index date)
5. Has a contraindication and is not eligible for treatment with brolucizumab according to the Beovu® (brolucizumab) Summary of Product Characteristics (SmPC) ("Beovu 120 mg/ml solution for injection in pre-filled syringe - Summary of Product Characteristics (SmPC)" 2020)
6. Any medical or psychological condition in the treating physician's opinion which may prevent the patient from participating in the study
7. Participating in a parallel interventional clinical study
8. Participating in a parallel non-interventional study (NIS) generating primary data for an anti- VEGF drug.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve the collection of data on adult patients with nAMD who have been newly initiated on brolucizumab at a participating NHS hospital
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of patients with absence of retinal fluid | Month 12
  Percentage (%) of patients with absence of retinal fluid (no Sub-retinal Fluid (SRF) and no Intra-retinal fluid (IRF) as documented in medical records by the treating physician in relation to OCT results)

SECONDARY OUTCOMES:
Percentage (%) of patients with absence of SRF | Month 3, month 6, month 12, month 24, month 36, month 48 and month 60
  Percentage (%) of patients without sub-retinal fluid (SRF) to be collected (fluid free)
Percentage (%) of patients with absence of IRF | Month 3, month 6, month 12, month 24, month 36, month 48 and month 60
  Percentage (%) of patients without intra-retinal fluid (IRF) to be collected (fluid-free)
Percentage (%) of patients with absence of sub-RPE fluid | Month 3, month 6, month 12, month 24, month 36, month 48 and month 60
  Percentage (%) of patients without sub-Retinal Pigment Epithelium fluid (sub-RPE) to be collected (fluid-free)
Percentage (%) of patients with absence of PED | Month 3, month 6, month 12, month 24, month 36, month 48 and month 60
  Percentage (%) of patients without retinal pigment epithelial detachment (PED) to be collected
Percentage (%) of patients with absence of retinal fluid | Month 3, month 6, month 12, month 24, month 36, month 48 and month 60
  Percentage (%) of patients without intra-retinal fluid (IRF), Sub-retinal Fluid (SRF) and sub-Retinal pigment epithelium (sub-RPE) fluid (fluid free) to be collected
CRT change from baseline | Baseline, month 3, month 6, month 12, month 24, month 36, month 48 and month 60
  measurement of Central Retinal Thickness (CRT) from baseline to be collected
CST change from baseline | Baseline, month 3, month 6, month 12, month 24, month 36, month 48 and month 60
  Measurement of Central Subfield Thickness (CST) from baseline to be collected
BCVA change from baseline | Baseline, month 3, month 6, month 12, month 24, month 36, month 48 and month 60
  Change in Best Corrected Visual Acuity (BCVA) from baseline to be corrected
Percentage (%) of patients with BCVA ≥70 ETDRS letters | Month 3, month 6, month 12, month 24, month 36, month 48 and month 60
  Percentage of patients with Best Corrected Visual Acuity (BCVA) ≥70 ETDRS letters to be collected
Total number of injections received | Up to 60 months
  Total number of injections received between Months 0 (index)-3, 4-6, 7-12, 0-12, 13-24, 25-36, 37-48, and 49-60
Duration of injection intervals per patient | Up to 60 months
  Duration of (all) injection intervals per patient during Months 0-6, 0-12, 13-24, 25-36, 37-48 and 49-60
Percentage (%) of patients with ≥3 brolucizumab injections | Month 3
  Percentage of patients completing the loading phase to be collected
Percentage (%) of patients who switch from brolucizumab to another anti-VEGF | Month 12, month 24, month 36, month 48 and month 60
  Percentage of patients who switch from brolucizumab to another anti-VEGF to be collected
Percentage (%) of patients that discontinue Brolucizumab therapy | Up to 60 months
  Percentage of patients that discontinue therapy to be collected
Percentage (%) of patients with IOI including RV and RVO | Up to 60 months
  Percentage of patients with Intraocular Inflammation (IOI) including Retinal vasculitis (RV) and Retinal vascular occlusion (RVO) to be collected
Percentage (%) of patients with disease control | Month 12 and month 24
  Percentage of patients with disease control, defined as absence of Intra-retinal fluid (IRF) and Sub-retinal Fluid (SRF), by the central reading center to be collected
Change in macular volume of IRF/SRF by central reading center | Baseline at Month 12
  Change in macular volume of IRF/SRF by central reading center according to type of fluid available at baseline. Macular volume will be quantified using a specialized validated AI algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United Kingdom (16):
  - Novartis Investigative Site, Peterborough, Cambridgeshire
  - Novartis Investigative Site, Abergele, Conwy
  - Novartis Investigative Site, Blackburn, Lancashire
  - Novartis Investigative Site, Uxbridge, London
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Barnsley
  - Novartis Investigative Site, Bedford
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Macclesfield
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Sunderland
  - Novartis Investigative Site, Warwick

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRTH258AGB02 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18238